CLINICAL TRIAL: NCT05470023
Title: Imaging-based Assessment of Oral Biofilm and Gingival Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Petra E. Wilder-Smith, Professor of Surgery and Director of Dentistry, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 881
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Plaque, Dental; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to different treatments.
Who Masked: Participant, Investigator
Masking Description: White tape over receptacle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Brushing with LivFresh Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with LivFresh Dental Gel with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Brushing with LivFree Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with LivFree Dental Gel with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Brushing with AIM Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with AIM Dental Gels with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Brushing with Crest Prohealth Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with Crest Prohealth Dental Gel with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Brushing with Parodontax Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with Parodontax Dental Gel with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Brushing with Colgate Total Dental Gel (Active Comparator): Subjects will brush twice daily for the study duration with Colgate Total Dental Gel with a standard Oral B ProFlexR toothbrush and will be trained in standard sulcular brushing technique. Subjects will brush their teeth two hours prior to each visit and refrain from eating from that time onwards until after their visit. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses
- Rinsing with Lumineux or Listerine Mouthwashes (Active Comparator): Subjects will be asked to rinse twice daily with 1 capful for 1 minute with Lumineux or Listerine Mouthwashes directly after brushing their teeth, while continuing with their usual oral hygiene protocol. Plaque levels, gingival inflammation, and sulcus bleeding will be recorded. A standardized periodontal probe will be used to measure pockets. Subjects will expectorate into a graduated cylinder for 5 minutes and their saliva production will be measured. Saliva will not be stored or analyzed in any way. Subjects will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images. These photos will not show the subject's face but will focus on the subject's mouth.
  Interventions: Other: OTC Toothpastes or Mouthrinses

INTERVENTIONS:
Other: OTC Toothpastes or Mouthrinses — OTC Toothpastes or mouthrinses used according to standard of care

SUMMARY:
The purpose of this research study is to develop a better way of measuring the health of patients' mouth using photographs and imaging software. The investigators will also study the specific effects of individual toothpastes and mouthwashes on oral health.

Participants who have volunteered to be in the study will be asked to use a toothpaste or over a period of 7 days to 6 months. The investigators will determine the participants' oral plaque levels, gum health, and saliva (spit) production with clinical exams as well as photographs of the participants' mouths. It is the hope of the study team to find better ways of assessing the health of patients' mouths and to identify whether gum health can be improved by specific toothpastes or mouthwashes.

DETAILED DESCRIPTION:
Participants will be asked whether they fulfill study inclusion/exclusion criteria. If recruited, they will be asked to sign the informed consent form. No professional dental cleaning will be performed before or during the trial in order to avoid the influence this would have on the data gathered. Participants will be randomly assigned to use one of the oral care products, which are all OTC products and will be used in the intended manner.

For toothpastes, participants will be asked to brush twice daily for the study duration with one of the following test dental gels: LivFresh Dental Gel (Livionex, Los Gatos, CA); LivFree Dental Gel (Los Gatos, CA); AIM (Church and Dwight, Ewing, NJ); Parodontax (GSK, Philadelphia, PA); Crest Prohealth (P&G, Cincinnati, OH); and Colgate Total (Colgate-Palmolive, New York, NY). A standard Oral B ProFlexR toothbrush will be provided to each volunteer, and participants will be trained in standard sulcular brushing technique. Participants will brush participants' teeth two hours prior to each visit and refrain from eating from that time onwards until after participants' visit. Participants allocated to mouthrinse use will continue with participants' usual oral hygiene protocol; additionally, the participants will be asked to rinse twice daily with 1 capful for 1 minute with the Lumineux Mouthrinse (Lumineux, Beverley Hills, CA) directly after brushing participants' teeth. Plaque levels (P.I.), gingival inflammation, and sulcus bleeding (mSBI) will be recorded.

A standardized periodontal probe will be used to measure pockets. Saliva production will be measured by asking participants to expectorate into a graduated cylinder for 5 minutes. Saliva will not be stored or analyzed in any way.

Volunteers will be photographed and evaluated on all study dates by the same blinded, pre-calibrated investigator. Photographs will be recorded using a standard dental intraoral camera, which only records intraoral images, thus automatically rendering the images unidentifiable with regard to each subject's facial appearance. These photos will not show the subject's face but will focus on the subject's mouth. Participants will be asked whether participants fulfill study inclusion/exclusion criteria inclusion/exclusion criteria.

Study duration will be 7 days or 1, 3, or 6 months. Each visit will last approximately 30 minutes. Initially, study duration will be 7 days as the investigators develop the imaging- based techniques. Once the techniques are finalized, study duration will be incrementally increased to 1 month, then 3 months, then 6 months to validate and refine the imaging-based techniques.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older
* In good general health

Exclusion Criteria:

* History of allergy or intolerance of oral hygiene products such as toothpastes and mouthrinses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Plaque level at Week 1 | 1 week
  Oral plaque will be measured using the gold standard plaque index (0-5; 0-best, 5 worst).
Plaque level at Month 1 | 1 month
  Oral plaque will be measured using the gold standard plaque index (0-5; 0-best, 5 worst).
Plaque level at Month 3 | 3 months
  Oral plaque will be measured using the gold standard plaque index (0-5; 0-best, 5 worst).
Plaque level at Month 6 | 6 months
  Oral plaque will be measured using the gold standard plaque index (0-5; 0-best, 5 worst).
Gingival health (gingival index) at Week 1 | 1 week
  Gingival health will be measured using the gold standard gingival index (0-3; 0-best, 3 worst).
Gingival health (gingival index) at Month 1 | 1 month
  Gingival health will be measured using the gold standard gingival index (0-3; 0-best, 3 worst).
Gingival health (gingival index) at Month 3 | 3 months
  Gingival health will be measured using the gold standard gingival index (0-3; 0-best, 3 worst).
Gingival health (gingival index) at Month 6 | 6 months
  Gingival health will be measured using the gold standard gingival index (0-3; 0-best, 3 worst).
Gingival health (sulcus bleeding index) at Week 1 | 1 week
  Gingival health will be measured using the gold standard modified sulcus bleeding index (0-3; 0-best, 3 worst).
Gingival health (sulcus bleeding index) at Month 1 | 1 month
  Gingival health will be measured using the gold standard modified sulcus bleeding index (0-3; 0-best, 3 worst).
Gingival health (sulcus bleeding index) at Month 3 | 3 months
  Gingival health will be measured using the gold standard modified sulcus bleeding index (0-3; 0-best, 3 worst).
Gingival health (sulcus bleeding index) at Month 6 | 6 months
  Gingival health will be measured using the gold standard modified sulcus bleeding index (0-3; 0-best, 3 worst).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Petra Wilder-Smith, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axelsson P, Lindhe J. The significance of maintenance care in the treatment of periodontal disease. J Clin Periodontol. 1981 Aug;8(4):281-94. doi: 10.1111/j.1600-051x.1981.tb02039.x. No abstract available. PMID 6947992
- [Background] Baek JH, Krasieva T, Tang S, Ahn Y, Kim CS, Vu D, Chen Z, Wilder-Smith P. Optical approach to the salivary pellicle. J Biomed Opt. 2009 Jul-Aug;14(4):044001. doi: 10.1117/1.3158994. PMID 19725713
- [Background] Colston BW Jr, Everett MJ, Da Silva LB, Otis LL, Stroeve P, Nathel H. Imaging of hard- and soft-tissue structure in the oral cavity by optical coherence tomography. Appl Opt. 1998 Jun 1;37(16):3582-5. doi: 10.1364/ao.37.003582. PMID 18273327
- [Background] Eke PI, Dye BA, Wei L, Thornton-Evans GO, Genco RJ; CDC Periodontal Disease Surveillance workgroup: James Beck (University of North Carolina, Chapel Hill, USA), Gordon Douglass (Past President, American Academy of Periodontology), Roy Page (University of Washin. Prevalence of periodontitis in adults in the United States: 2009 and 2010. J Dent Res. 2012 Oct;91(10):914-20. doi: 10.1177/0022034512457373. Epub 2012 Aug 30. PMID 22935673
- [Background] Haffajee AD, Socransky SS. Microbial etiological agents of destructive periodontal diseases. Periodontol 2000. 1994 Jun;5:78-111. doi: 10.1111/j.1600-0757.1994.tb00020.x. No abstract available. PMID 9673164
- [Background] Llena-Puy C. The role of saliva in maintaining oral health and as an aid to diagnosis. Med Oral Patol Oral Cir Bucal. 2006 Aug;11(5):E449-55. English, Spanish. PMID 16878065
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Madlena M, Banoczy J, Gotz G, Marton S, Kaan M Jr, Nagy G. Effects of amine and stannous fluorides on plaque accumulation and gingival health in orthodontic patients treated with fixed appliances: a pilot study. Oral Health Dent Manag. 2012 Jun;11(2):57-61. PMID 22692271
- [Background] Morris AJ, Steele J, White DA. The oral cleanliness and periodontal health of UK adults in 1998. Br Dent J. 2001 Aug 25;191(4):186-92. doi: 10.1038/sj.bdj.4801135. PMID 11551090
- [Background] Nogueira-Filho GR, Toledo S, Cury JA. Effect of 3 dentifrices containing triclosan and various additives. An experimental gingivitis study. J Clin Periodontol. 2000 Jul;27(7):494-8. doi: 10.1034/j.1600-051x.2000.027007494.x. PMID 10914890
- [Background] Theilade E, Wright WH, Jensen SB, Loe H. Experimental gingivitis in man. II. A longitudinal clinical and bacteriological investigation. J Periodontal Res. 1966;1:1-13. doi: 10.1111/j.1600-0765.1966.tb01842.x. No abstract available. PMID 4224181
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] van der Weijden GA, Hioe KP. A systematic review of the effectiveness of self-performed mechanical plaque removal in adults with gingivitis using a manual toothbrush. J Clin Periodontol. 2005;32 Suppl 6:214-28. doi: 10.1111/j.1600-051X.2005.00795.x. PMID 16128840
- [Background] Yates R, Jenkins S, Newcombe R, Wade W, Moran J, Addy M. A 6-month home usage trial of a 1% chlorhexidine toothpaste (1). Effects on plaque, gingivitis, calculus and toothstaining. J Clin Periodontol. 1993 Feb;20(2):130-8. doi: 10.1111/j.1600-051x.1993.tb00327.x. PMID 8436632